CLINICAL TRIAL: NCT04367363
Title: Tracking WhatsApp Behaviors During a Crisis: A Longitudinal Observation of Messaging Activities During the COVID-19 Pandemic
Brief Title: Social Media and COVID-19
Status: Completed | Type: Observational
Sponsor: Jean Liu (Other)
Responsible Party: Sponsor-Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Organization: Yale-NUS College (Other)
Other Study IDs: 2020-CERC-001B
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus; Depression; Anxiety; Stress
Keywords: Social Media; Misinformation; COVID-19
MeSH Terms: conditions — Coronavirus Infections; Depression; Anxiety Disorders; Communication; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: We plan to recruit a representative sample of the Singapore population.
  Interventions: Behavioral: Social media & news consumption

INTERVENTIONS:
Behavioral: Social media & news consumption — Daily reports of social media use and consumption, including reports on receiving and disseminating news articles related to the COVID-19 situation (e.g., how many messaging groups shared news on the outbreak, how many items related to the outbreak they forwarded to others, etc).

SUMMARY:
In this protocol, we seek to examine the role of popular messaging platform WhatsApp in information spread during a crisis. As there have been few global crises in the last decade (coinciding with the rise of social media), the role of private messaging platforms such as WhatsApp during crisis contexts remains understudied. During the current COVID-19 global health crisis, we undertook this study to: (1) characterize the nature of WhatsApp use during crises, (2) characterize the profiles of WhatsApp users (3) understand how WhatsApp usage links to well-being (fear and thoughts about COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years
* Has stayed in Singapore for at least 2 years
* Has a WhatsApp account that can be used for the research study

Exclusion Criteria:

* Below 21 years
* Has stayed in Singapore for less than 2 years
* Does not have a WhatsApp account that can be used for the research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative sample of the Singapore population
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
WhatsApp usage | 1 week, starting from date after baseline survey completion
  Participants were asked a series of questions daily related to their WhatsApp usage behaviors - in particular, their message-forwarding, personal chat and group chat behaviors.
Changes in fear with regards the COVID-19 situation across 1 week | 1 week, starting from date after baseline survey completion
  1 item each day on fear specifically of the COVID-19 situation (measured on a 4 point scale: min = 1, max = 4; higher scores indicating greater fear about the outbreak).
Changes in amount of thinking about the COVID-19 situation across 1 week | 1 week, starting from date after initial survey completion
  1 item each day on how much they thought about the outbreak that day (measured on a 5 point scale: min = 1, max = 5; higher scores indicating more thinking about the outbreak).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liu, PhD, Principal Investigator — Yale-NUS College
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the Institutional Review Board, data cannot be shared.

REFERENCES:
- [Derived] Tan EY, Wee RR, Saw YE, Heng KJ, Chin JW, Tong EM, Liu JC. Tracking Private WhatsApp Discourse About COVID-19 in Singapore: Longitudinal Infodemiology Study. J Med Internet Res. 2021 Dec 23;23(12):e34218. doi: 10.2196/34218. PMID 34881720